CLINICAL TRIAL: NCT04627415
Title: Early Intervention for Young Children At-Risk for ADHD: Evaluating Efficacy and Delivery Format for Behavioral Parent Education
Brief Title: Project PEAK: Early Intervention for ADHD
Acronym: PEAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, George DuPaul, Associate Dean for Research; Professor of School Psychology, Lehigh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IES: R324A200010
Record Dates: First submitted 2020-10-27; First posted 2020-11-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit Hyperactivity Disorder; Parent-Child Relations; Child Behavior; Parenting
Keywords: ADHD; Behavioral Parent Training; Early Intervention; Preschool
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Face to Face Treatment (Experimental): The F2F version of PEAK contains 10 BPE sessions (1.5 hours each). Session content includes: 1) Introduction to ADHD, 2) Attending, Rewards and Ignoring, 3) General Behavior Management Strategies, 4) Problem-Solving Approach, 5) Preventive Intervention, 6) Instructive Interventions, 7) Response Strategies, 8) Extending What Works to Community Settings, 9) Promoting Early Reading and Math Skills, and 10) Effective Communication Strategies. Each session contains didactic instruction and activities designed to enhance engagement. Sessions include video examples and interactive activities. Weekly homework is assigned for strategy practice. At the start of the following session, the leader checks in with families on the use of the chosen strategy. The session leader praises successes and troubleshoots challenges. The intervention also includes optimistic training which aims to identify/improve pessimistic thinking patterns that parents have about their parenting and child's behaviors.
  Interventions: Behavioral: Promoting Engagement with ADHD Pre-Kindergarteners
- Online Treatment (Experimental): For the online version of the program, in addition to content regarding an overview of ADHD, the initial session consists of brief video clips demonstrating how to access PEAK sessions on the Internet, and an orientation to online content (e.g., handouts, interactive chat sessions, research team contact links). Prior to the session, parents are provided with password-protected individual access codes. Similar to the F2F program, check-ins are provided weekly via each parent's preferred mode of communication (i.e., text, internet, phone) to query strategies implemented, praise success, and troubleshoot alternative strategies. Parents in the online condition will also receive supplemental optimistic training to improve pessimistic thinking patterns about their child and parenting.
  Interventions: Behavioral: Promoting Engagement with ADHD Pre-Kindergarteners
- Waitlist Control (Other): The comparison condition is a waitlist control group that will receive no intervention throughout the intervention timeframe. Instead, participants will receive wellness information about typical child development and constructs unrelated to the intervention content. Subsequent to the 12-month follow-up assessment, they will be provided access to the online version of the program. To encourage ongoing participation in the absence of services, parents will be informed that, at the end of the intervention timeframe, they will receive support (i.e., weekly contact to answer questions) while they complete the online program.
  Interventions: Behavioral: Promoting Engagement with ADHD Pre-Kindergarteners

INTERVENTIONS:
Behavioral: Promoting Engagement with ADHD Pre-Kindergarteners — Optimism Training includes the following strategies: 1) Identifying situations and associations 2) Determining consequences of beliefs 3) Use distractions to interrupt negative thinking 4) dispute current thinking 5) substitute positive, productive thoughts 6) practice skills to recognize/modify self-talk 7) Maintain positive changes in self-talk
  Other Names: PEAK; Optimism Training

SUMMARY:
Parent education is an effective and relatively cost efficient approach for reducing child behavior problems. Research, however, suggests that the effectiveness of parent education is mitigated by parent attendance and parent implementation of intervention strategies. That is, low attendance at parent education sessions is associated with limited intervention effects. Therefore, it is critical to identify strategies to enhance parent engagement. A previous pilot randomized controlled trial of a parent education program (Behavioral Parent Education; BPE, specifically Promoting Engagement for ADHD pre-Kindergartners [PEAK]), found that both face-to-face (F2F) and online BPE resulted in high levels of parent engagement and child behavior improvements. However, results need to be replicated in a full scale efficacy trial with a larger, diverse sample to provide more reliable estimates of relative effect sizes for parent and child outcomes and to evaluate the extent to which parent and child behavior changes are maintained after BPE has ended. In the current randomized controlled trial, the investigators intend to apply What Works Clearinghouse group design standards to examine the efficacy of two forms of delivery of BPE (F2F and online) relative to a wait-list control condition in a sample of 180, 3- to 5-year old children with clinically significant symptoms of ADHD. The objective is to: (a) extend findings from the pilot investigation to a large, diverse sample; (b) examine maintenance of effects; (c) identify moderators and mediators of treatment outcome, especially the degree to which these may differ for F2F vs. online treatment delivery; and (d) assess cost and cost-effectiveness of the two PEAK delivery formats.

DETAILED DESCRIPTION:
PEAK addresses potential barriers to treatment access and engagement in at least four ways. First, the 10 sessions require fewer hours to complete relative to typical BPE programs. Second, PEAK content and process was developed with extensive input from primary stakeholders (i.e., parents of young children with ADHD). The iterative process used in the Development grant provided critical parental input regarding revision to maximize engagement. Third, the availability of online treatment delivery allows greater flexibility relative to F2F delivery in terms of time and location of completing BPE sessions. This should increase access for families with limited resources (e.g., transportation) or constrained schedules. Finally, online delivery may be less costly to access given need for fewer resources (e.g., space, child care), although relative cost-effectiveness will be explored in greater detail in the proposed project.

Intervention Components. Both the F2F and online versions of PEAK contain 10 scripted BPE sessions that last approximately 1.5 hours. Session content includes: 1) Introduction to ADHD, 2) Attending, Rewards and Ignoring, 3) General Behavior Management Strategies, 4) Problem-Solving Approach, 5) Preventive Intervention, 6) Instructive Interventions, 7) Response Strategies, 8) Extending What Works to Community Settings, 9) Promoting Early Reading and Math Skills, and 10) Effective Communication Strategies. Supplemental Optimism Training will also be included to help parents identify/improve pessimistic thoughts about their parenting and their child's behavior. Each session contains didactic instruction interspersed with activities designed to enhance parent engagement. Sessions include video examples and interactive activities, such as role-play, group discussion for F2F, and check-in questions for online. Weekly homework activities are assigned for strategy practice. For example, parents choose one strategy (e.g., transitional warning, timer, choice) discussed during the session to implement at home. At the start of the following session, the session leader checks in with families on the use of the chosen strategy. The session leader praises successes and troubleshoots where strategy implementation went awry, suggesting alternative strategies or implementation approaches.

For the online version of the program, parents are provided with password- protected individual access codes to the online PEAK program. Check-ins are provided weekly via each parent's preferred mode of communication (i.e., text, internet, phone) to query strategies implemented, praise success, and troubleshoot alternative strategies.

Both the F2F and online versions of PEAK address many of the inner and outer contextual variables, particularly those that are malleable. For example, streamlined and/or online BPE may ease access challenges related to single parent status, inflexible treatment hours/location, or perceived stigma associated with obtaining mental health treatment. Program content is designed to enhance perceived sense of parenting efficacy through ongoing feedback from PEAK staff regarding use of strategies. Similarly, content is designed to provide parents with accurate attributions for child behavior difficulties in the context of understanding ADHD as well as environmental factors impacting behavior (e.g., antecedents, consequences). PEAK also includes content designed to help parents communicate and collaborate with teachers and school personnel.

Process and Materials. The F2F program is fully manualized, with each session consisting of slides, scripted presentation notes, and activities. Advanced graduate students in School Psychology or Special Education who have completed courses in Consultation and Positive Behavior Support serve as Session Leaders. To assure high quality delivery, the Principal Investigator (PI) or co-PI attends the first session and provides feedback to the Session Leader. All sessions are audiorecorded and the PI or co-PI listens to each recorded session weekly and completes a fidelity checklist. Weekly feedback is provided to the Session Leader regarding strengths and areas for improvement.

The online format is fully developed and ready for parent use. It consists of identical content, handouts, and practice activities to the F2F version. A Web Designer with expertise in technology is designated to address technical difficulties.

Intervention Context. The PEAK program is intended for parents of young children, ages 3-5, at-risk for ADHD. Children had to have met Diagnostic and Statistical Manual-5 criteria for one of the three presentations of ADHD based on clinical interview, parent/teacher behavior ratings (90th percentile). However, for future use, the investigators anticipate the program being equally (if not more) effective with children with less severe symptoms. Children were excluded who had diagnoses of autism spectrum disorder (ASD), pervasive developmental disorder, intellectual disability, neurological damage, or significant motor or physical impairments.

A variety of care providers participated in the intervention and will be end users, including biological parents, stepparents, foster parents, significant others, and grandparents with custody of their grandchildren. The only restriction was that at least one English-speaking parent needed to participate because the program and assessments are in English. In addition, parents had to have an electronic device with Internet access (assessed prior to randomization) and express willingness to attend F2F meetings or complete online sessions.

Theory of Change. PEAK was designed to address two target areas that are specifically problematic for young children at-risk for ADHD: poor parent-child interactions and difficulty with pre-academic skills. the investigators have sequenced sessions such that skills that have a theoretical overlap across components are taught first. Specifically, skills that comprise desirable parent-child interactions (e.g., providing praise, following through, offering constructive feedback) should be employed when engaged in activities to enhance pre-academic skills (taught in the last session). At the same time, there are strategies distinct to each intervention area. For instance, pre-academic readiness requires that parents engage in specific pre-academic activities.

The purpose of the proposed randomized control trial (RCT) is to apply What Works Clearinghouse group design standards to examine the initial efficacy of two forms of delivery of streamlined BPE (F2F and online) relative to a wait-list control condition in a sample of 3- to 5-year old children with clinically significant symptoms of ADHD. The objective is to: (a) extend findings from the pilot investigation to a large, diverse sample; (b) examine maintenance of effects; (c) identify moderators and mediators of treatment outcome, especially the degree to which these may differ for F2F vs. online treatment delivery; and (d) assess cost and cost-effectiveness of the two PEAK delivery formats. The specific aims are described below.

Aim 1: Examine the immediate post-treatment effects of F2F and online BPE relative to a wait-list control (WLC) condition on parent knowledge of and fidelity with intervention strategies, parent acceptability of training procedures and interventions, child early academic skills, and child and parent behavior for families of young children at-risk for ADHD.

Based on the pilot RCT findings, the investigators hypothesize that F2F and online BPE will lead to significantly greater improvement at post-treatment in parent knowledge of and fidelity with intervention strategies as well as child and parent behavior relative to WLC. The investigators do not expect that the two BPE conditions will differ with respect to these outcomes. Also based on the pilot RCT, the investigators expect treatment acceptability to be in the moderate to high range for both active treatment conditions with significantly higher ratings for F2F intervention. Finally, the investigators hypothesize small but statistically significant gains in child early academic skills for the F2F and online conditions relative to WLC, with no difference between active treatment conditions.

Aim 2: Evaluate the degree to which post-treatment effects maintain at 6-month intervals for up to 2 years and whether maintenance of effects differs between groups for up to 1 year for all participants and up to 2 years for those controls who do not participate in treatment.

Based on prior studies of BPE, the investigators expect post-treatment effects on child and parent behavior to maintain across the up to 2-year follow-up period with F2F and online BPE continuing to differ from WLC and no differences between F2F and online BPE.

Aim 3: Identify possible moderators (i.e., parent session completion, parent income, education, marital status, and parent ADHD symptoms) and mediators (i.e., parent knowledge, fidelity, and stress) of treatment-induced changes in child behavior and early academic skills as a function of BPE and examine whether moderators/mediators differ as a function of BPE delivery format. This aim will involve identifying variables that predict differential response to F2F vs. online BPE delivery formats (i.e., what variables predict which families will benefit most from one delivery format vs. the other).

Based on prior BPE studies, the investigators hypothesize that treatment effects will be greater for participants who complete all sessions and parents with less severe ADHD symptoms. Based on the pilot RCT findings, the investigators hypothesize that BPE effects on child behavior will be mediated by increases in parent knowledge and intervention fidelity along with concomitant reductions in parent stress. Because no prior studies have examined differential response to F2F versus online BPE, the examination of predictors of differential response to treatment delivery format is exploratory; thus, the investigators have no specific hypotheses in this area.

Aim 4: Identify costs associated with F2F and online BPE as well as compare cost-effectiveness between the two delivery formats.

ELIGIBILITY:
Inclusion Criteria:

* 3- to 5.11-year old children with clinically significant symptoms of ADHD.
* Children had to have met DSM-5 criteria for one of the three presentations of ADHD based on clinical interview and parent and teacher behavior ratings, including parent and teacher report of elevated levels of impairment at home and school (i.e., score greater than 90th percentile on one or more Conners Early Childhood Rating Scale subscales relevant to ADHD).

Exclusion Criteria:

* A diagnoses of autism spectrum disorder (ASD), pervasive developmental disorder, intellectual disability, neurological damage, or significant motor or physical impairments.
* Children needed to be enrolled in a pre-school or day care setting at least 2 days a week unless otherwise unable to enroll (e.g. behavioral problems, lack of services for unrelated disability) in order to establish the presence of symptoms across two settings.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-Treatment Effects (Parent): Intervention Strategies | 10 weeks
  To assess changes in intervention strategy use the test of parent knowledge (R= 0-15) and parent fidelity (R= 0-9) form will be used (higher scores = better outcomes).
Post-Treatment Effects (Parent): Behavior | 10 weeks
  To assess changes in parent behavior the Parenting Young Children (R= 22-154; higher scores = better outcomes), the DPICS and RPC (higher scores on negative codes = worse outcomes and higher scores on positive codes = better outcomes)
Post-Treatment Effects (Parent): Acceptability | 10 weeks
  To assess treatment acceptability the Intervention rating profile-15 (R= 15-90; higher scores = better outcomes) will be used.
Post-Treatment Effects (Parent): Stress | 10 weeks
  To assess chases in parenting stress, The Parenting Stress Inventory-4 (R=36-180; higher scores = worse outcomes) will be used.
Post-Treatment Effects (Parent): Optimism | 10 weeks
  To examine parental optimism post-treatment group comparisons, the Parental Attribution Measure (R= 0-12; higher scores = worse outcomes); The Family Empowerment Scale-Competence (R= 8-40; higher scores = better outcomes), and the Questionnaire on Resources and Stress-Pessimism (R=0-11; higher scores = worse outcomes) will be used.
Post-Treatment Effects (Child): Academics | 10 weeks
  To assess changes in child early academic skills the Individual Growth and Development Indicators of Early Learning (R=2.16-36.61; higher scores indicate better outcomes) will be used.
Post-Treatment Effects (Child): Behavior | 10 weeks
  To examine changes in child behavior the Conners-EC Rating Scale (R=0-100, higher scores indicate worse outcomes except for the developmental milestones)
Post-Treatment Effects (Child): Behavior Observations | 10 weeks
  To examine changes in child behavior the Dyadic Parent-Child Interactive Coding System-Revised (DPICS) and Relationship Process Code-2 (RPC) (higher scores on negative codes = worse outcomes and higher scores on positive codes = better outcomes)
Post-Treatment Effects (Child): Self Regulation | 10 weeks
  To examine changes in child self-regulation, the Head-Toes-Knees-Shoulders-Task (R=0-16; higher scores indicate better outcomes)
Post-Treatment Effects (Child): Bedtime Behaviors | 10 weeks
  To examine changes in child bedtime behaviors behaviors the Children's Sleep-Wake Scale-GTBS (R=5-30; higher scores indicate better outcomes).
Post-Treatment Effects (Child): Social Behaviors | 10 weeks
  To assess changes in child social behaviors the Adaptive Social Behavior Inventory (R=30-90; higher scores indicate worse outcomes) will be used
Post-Treatment Effects (Child): Social Behaviors | 2 years
  To assess maintenance in child social behaviors the Adaptive Social Behavior Inventory (R=30-90; higher scores indicate worse outcomes) will be used
Maintenance (Child): Behavior Observations | 2 years
  To examine maintenance in child behavior the Dyadic Parent-Child Interactive Coding System-Revised (DPICS) and Relationship Process Code-2 (RPC) (higher scores on negative codes = worse outcomes and higher scores on positive codes = better outcomes)
Maintenance (Child): Self Regulation | 2 years
  To examine maintenance in child self-regulation, the Head-Toes-Knees-Shoulders-Task (R=0-16; higher scores indicate better outcomes)
Maintenance (Child): Bedtime Behaviors | 2 years
  To examine maintenance in child bedtime behaviors behaviors the Children's Sleep-Wake Scale-GTBS (R=5-30; higher scores indicate better outcomes).
Maintenance (Parent): Acceptability | 2 years
  To assess maintenance of treatment acceptability the Intervention rating profile-15 (R= 15-90; higher scores = better outcomes) will be used.
Maintenance (Parent): Behavior | 2 years
  To assess maintenance in parent behavior the Parenting Young Children (R= 22-154; higher scores = better outcomes), the DPICS and RPC (higher scores on negative codes = worse outcomes and higher scores on positive codes = better outcomes)
Maintenance (Parent): Intervention Strategies | 2 years
  To assess maintenance in intervention strategy use the test of parent knowledge (R= 0-15) and parent fidelity (R= 0-9) form will be used (higher scores = better outcomes).
Maintenance (Parent): Stress | 2 years
  To assess maintenance in parenting stress, The Parenting Stress Inventory-4 (R=36-180; higher scores = worse outcomes) will be used.
Maintenance (Parent): Optimism | 2 years
  To examine maintenance in parental optimism, the Parental Attribution Measure (R= 0-12; higher scores = worse outcomes), The Family Empowerment Scale-Competence (R= 8-40; higher scores = better outcomes), and the Questionnaire on Resources and Stress-Pessimism (R=0-11; higher scores = worse outcomes) will be used.
Mediators and Moderators (Parent): Session Completion | 2 years
  To examine parent session completion, a frequency count will be used (higher scores= better outcomes).
Mediators and Moderators (Parent): Demographics | 2 years
  To assess parent income, education, and marital status the Parent Demographic Information form will be used.
Mediators and Moderators (Parent): ADHD Symptoms | 2 years
  Parent ADHD symptoms will be assessed using the Adult Investigator Symptom Rating Scale (R=18-90; higher scores= worse outcomes).
Mediators and Moderators (Parent): Parent Strategies | 2 years
  The test of parent knowledge (R= 0-15) and fidelity checklist (R= 0-9) (higher scores = better outcomes) will be used.
Mediators and Moderators (Parent): Stress | 2 years
  To assess parent stress, the Parenting Stress Inventory (PSI) will be used (R=36-180; higher scores = worse outcomes).
Mediators and Moderators (Parent): Media | 2 years
  Parent media use preference the Media and Technology Usage and Attitudes Scale (MTUAS) (R=45-506; higher scores = better outcomes) will be used.
Mediators and Moderators (Child) | 2 years
  To assess child self regulation the Head-Toes-Knees-Shoulders-Task (HTSK) will be used (R=0-16; higher scores indicate better outcomes).
Cost-Effectiveness (money): Face-to-face | 5 years
  Investigators will determine costs of the F2F program using the ingredients method by documenting cost of: (a) session leader, based on required minimal qualifications and salary for position ($); (b) space to run sessions ($ to rent out space) (d) food provided during session ($ for cost of food); (c) childcare provided during session ($ for childcare per hour); and (d) transportation, calculated by number of families needing transportation divided by total number of families (multiplied by average miles round trip x average Uber fare). Investigators will review effectiveness metrics by stratifying participants based on their characteristics (parent education level, socioeconomic index, ADHD medication status) prior to the intervention. Investigators will compare cost against effectiveness using Incremental Cost-Effectiveness Ratio (ICER).
Cost-Effectiveness (time): Face-to-face | 5 years
  Investigators will determine costs of the F2F program using the ingredients method by documenting time of: Individual contact hours by provider with minimal qualifications to support families between sessions (calculated as minutes of contact across efficacy trial divided by number of families). Investigators will review effectiveness metrics by stratifying participants based on their characteristics (parent education level, socioeconomic index, ADHD medication status) prior to the intervention. Investigators will compare cost against effectiveness using Incremental Cost-Effectiveness Ratio (ICER).
Cost-Effectiveness (time): Online | 5 years
  For the online program, we will determine costs (in time) of (a) individual contact hours by provider with minimal qualifications to support families between sessions, calculated as minutes of contact across efficacy trial divided by number of families; (b) technology support for families, as provided by technology expert with minimal qualifications and calculated as minutes spent supporting families with user challenges divided by total number of families in efficacy trial; and (c) technology support on creator end, as provided by technology expert with minimal qualifications and calculated as minutes spent. Investigators will review effectiveness metrics by stratifying participants based on their characteristics (parent education level, socioeconomic index, ADHD medication status) prior to the intervention. Investigators will compare cost against effectiveness using Incremental Cost-Effectiveness Ratio (ICER).
Cost-Effectiveness (money): Online | 5 years
  For the online program, we will determine costs of purchase of phone and data plan for approximately 10% of families without internet access. Investigators will review effectiveness metrics by stratifying participants based on their characteristics (parent education level, socioeconomic index, ADHD medication status) prior to the intervention. Investigators will compare cost against effectiveness using Incremental Cost-Effectiveness Ratio (ICER).

CONTACTS AND LOCATIONS:
Overall Officials: George J DuPaul, Ph.D., Principal Investigator — Lehigh University; Lee Kern, Ph.D., Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States